CLINICAL TRIAL: NCT04365946
Title: Microbiome Analysis in Patients With Gastric Intestinal Metaplasia and in Patients With Gastric Cancer and Correlation With the Subtypes of the Lesions
Brief Title: Microbiome Analysis in Gastric Intestinal Metaplasia and in Gastric Cancer and Subtypes Correlation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Ioannina (Other)
Collaborators: University of Ioannina (Other)
Responsible Party: Principal Investigator, George Pappas-Gogos, George Pappas-Gogos, Principal Investigator, University Hospital, Ioannina
Other Study IDs: 1
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Gastric Intestinal Metaplasia; Gastric Cancer; Microbiome
Keywords: Gastric intestinal metaplasia; Gastric cancer; Subtypes; Microbiome
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Complete type: Patients with complete-type intestinal metaplasia
  Interventions: Procedure: Gastroscopy
- Incomplete type: Patients with incomplete-type intestinal metaplasia
  Interventions: Procedure: Gastroscopy
- Controls: Healthy subjects
  Interventions: Procedure: Gastroscopy

INTERVENTIONS:
Procedure: Gastroscopy — Upper GI endoscopy and biopsy

SUMMARY:
The aim of the study will be to analyze the microbiome in the blood and stomach in patients with intestinal metaplasia (IM) and / or gastric cancer (GC). As far as IM is concerned, it has been found that the incomplete type is related to GC mainly intestinal-type. Studies show differences in the microbiome in patients with IM and in patients with GC, but do not specify whether these differences are related to histological types.

Our intention is to further analyze the microbiome based on histological types. Most studies on stomach cancer have focused on the microbiota of gastric microbiota. Recent data have shown that the microbiome of the small intestine, especially the mucosa, can play a key role in the condition of the gastrointestinal tract. Disturbance of the microbiome of the small intestine has been found in celiac disease, chronic liver disease, diabetes and irritable bowel syndrome. However, information on the role of the microbiome in IM remains limited.

DETAILED DESCRIPTION:
Review of research area Intestinal metaplasia of the stomach (IM) is generally considered a precancerous lesion and is associated with a small increase in the risk of developing gastric cancer (GC). Endoscopic monitoring has been proposed to control the risk of endangered populations. However, due to the lower incidence of GC in the United States and other Western countries, there is no specific monitoring protocol. In general, there are no widely accepted guidelines for IM management. Recently, the European Endoscopic Society as well as other European academic companies have developed documented guidelines for the management of patients with IM.

These guidelines emphasize the increased risk of cancer in patients with gastric atrophy and IM and the need for staging in cases of high-grade dysplasia. Risk factors for IM include Helicobacter pylori infection, high NaCl intake, smoking, alcohol consumption and chronic biliary reflux.

The development of intestinal-type gastric carcinoma occurs in four stages: non-atrophic gastritis, multifocal atrophic gastritis, IM, and dysplasia. The IM of the gastric cardia and the Barrett's esophagus differ in the risk of malignancy. Elevated serum pepsinogen levels have been suggested as an indicator of extensive gastric atrophy. Currently, there are no reliable markers of gastric dysplasia or gastric cancer.

Based on the available data, it appears that the IM of the gastric cardia is a possible precursor to the development of intestinal-type carcinoma of the stomach. It has been found that 45% of patients with gastric carcinoma had residual IM, supporting the idea that IM is a particularly important precursor to its development. Histologically, the IM may be complete or incomplete. Complete (type I) intestinal metaplasia is defined by the mucosa of the small intestinal type with mature absorbent cells, cell cups, and a brush-like outline. Incomplete intestinal metaplasia (type II) secretes cialomycin and is similar to colonic epithelium with columns of "intermediate" cells at various stages of differentiation, irregular mucosal droplets and the absence of a "brush" limit. The highest risk of gastric cancer is associated with incomplete and / or extensive IM.

Recent studies show that microbial changes are related to the histological stages of gastric oncogenesis. Chronic H. pylori infection can cause inflammation of the mucosa and cause histological changes. It is also recognized as an important risk factor for GC. However, only 3% of patients infected with H. pylori develop GC. In addition, H. pylori has been found to be usually undetectable in GC samples. These studies suggest that H. pylori infection may only be an early event for the gastric mucosa, which will undergo further oncogenic changes and indicate the possible role of mucosal microbes, with the exception of H. pylori in the gastric carcinoma.

The dominant germ type in the gastric mucosa was found to be protein-secreted bacteria, in both H. pylori negative and positive for H. pylori samples. Two previous studies have shown that the microbial count in IM patients was found to be partially overlapped with the group of gastritis and cancer among patients with H. pylori infection. Li et al (2017) found that the microbial amount in gastritis samples overlapped mostly with that of IM samples. In contrast, the microflora of patients with IM and GC had significantly lower microbial richness, while the biodiversity of the microbiology of patients with overt gastritis (EG), chronic gastritis (CG) and IM was similar in total, with the exception of those with GC. These conflicting results suggest that IM may be the key point in microbial change and that there may be other qualitative factors involved in gastric oncogenesis, especially in patients with IM.

Research subject and objectives The study will be performed on patients undergoing gastroscopy who have IM and / or GC findings. In patients with IM, the microbiome will be analyzed and correlated with the type of IM (complete-incomplete). The same will be done for patients with GC (intestinal-type cancer).

Thematic area The aim of the study will be to analyze the microbiome in the blood and stomach in patients with intestinal metaplasia (IM) and / or gastric cancer (GC). As far as IM is concerned, it has been found that the incomplete type is related to GC mainly intestinal-type. Studies show differences in the microbiome in patients with IM and in patients with GC, but do not specify whether these differences are related to histological types.

Our intention is to further analyze the microbiome based on histological types. Most studies on stomach cancer have focused on the microbiota of gastric microbiota. Recent data have shown that the microbiome of the small intestine, especially the mucosa, can play a key role in the condition of the gastrointestinal tract. Disturbance of the microbiome of the small intestine has been found in celiac disease, chronic liver disease, diabetes and irritable bowel syndrome. However, information on the role of the microbiome in IM remains limited.

Keywords Gastric intestinal metaplasia, Complete Type, Incomplete Type, Gastric Cancer, Microbiome

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric intestinal metaplasia and/or gastric cancer
* Healthy controls

Exclusion Criteria:

* Metabolic syndrome and its components
* IBD
* Autoimmune diseases
* Otherwise tumours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gastric intestinal metaplasia and/or gastric cancer, and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Analysis of microbiome in subtypes of intestinal metaplasia and gastric cancer | Through study completion, an average of 1 year.
  Microbiome analysis with complete and incomplete type of intestinal metaplasia and subtypes of gastric cancer
Analysis of microbiome in subtypes of intestinal metaplasia and gastric cancer | Through study completion, an average of 1 year.
  Microbiome correlation with complete and incomplete type of intestinal metaplasia and subtypes of gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Vlachos, Prof, Study Director — University of Ioannina; George Pappas-Gogos, Dr, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2021-2023
Access Criteria: Researchers who would access data, statistics and results of this study in order to perform similar studies

REFERENCES:
- [Background] Gao JJ, Zhang Y, Gerhard M, Mejias-Luque R, Zhang L, Vieth M, Ma JL, Bajbouj M, Suchanek S, Liu WD, Ulm K, Quante M, Li ZX, Zhou T, Schmid R, Classen M, Li WQ, You WC, Pan KF. Association Between Gut Microbiota and Helicobacter pylori-Related Gastric Lesions in a High-Risk Population of Gastric Cancer. Front Cell Infect Microbiol. 2018 Jun 19;8:202. doi: 10.3389/fcimb.2018.00202. eCollection 2018. PMID 29971220
- [Background] Liu X, Shao L, Liu X, Ji F, Mei Y, Cheng Y, Liu F, Yan C, Li L, Ling Z. Alterations of gastric mucosal microbiota across different stomach microhabitats in a cohort of 276 patients with gastric cancer. EBioMedicine. 2019 Feb;40:336-348. doi: 10.1016/j.ebiom.2018.12.034. Epub 2018 Dec 21. PMID 30584008
- [Background] Wang L, Zhou J, Xin Y, Geng C, Tian Z, Yu X, Dong Q. Bacterial overgrowth and diversification of microbiota in gastric cancer. Eur J Gastroenterol Hepatol. 2016 Mar;28(3):261-6. doi: 10.1097/MEG.0000000000000542. PMID 26657453
- [Background] Gong J, Li L, Zuo X, Li Y. Change of the duodenal mucosa-associated microbiota is related to intestinal metaplasia. BMC Microbiol. 2019 Dec 9;19(1):275. doi: 10.1186/s12866-019-1666-5. PMID 31815623
- [Background] Eun CS, Kim BK, Han DS, Kim SY, Kim KM, Choi BY, Song KS, Kim YS, Kim JF. Differences in gastric mucosal microbiota profiling in patients with chronic gastritis, intestinal metaplasia, and gastric cancer using pyrosequencing methods. Helicobacter. 2014 Dec;19(6):407-16. doi: 10.1111/hel.12145. Epub 2014 Jul 23. PMID 25052961
- [Background] Park CH, Lee AR, Lee YR, Eun CS, Lee SK, Han DS. Evaluation of gastric microbiome and metagenomic function in patients with intestinal metaplasia using 16S rRNA gene sequencing. Helicobacter. 2019 Feb;24(1):e12547. doi: 10.1111/hel.12547. Epub 2018 Nov 15. PMID 30440093
- [Background] Hsieh YY, Tung SY, Pan HY, Yen CW, Xu HW, Lin YJ, Deng YF, Hsu WT, Wu CS, Li C. Increased Abundance of Clostridium and Fusobacterium in Gastric Microbiota of Patients with Gastric Cancer in Taiwan. Sci Rep. 2018 Jan 9;8(1):158. doi: 10.1038/s41598-017-18596-0. PMID 29317709
- [Background] Park CH, Lee JG, Lee AR, Eun CS, Han DS. Network construction of gastric microbiome and organization of microbial modules associated with gastric carcinogenesis. Sci Rep. 2019 Aug 27;9(1):12444. doi: 10.1038/s41598-019-48925-4. PMID 31455798
- [Background] Jencks DS, Adam JD, Borum ML, Koh JM, Stephen S, Doman DB. Overview of Current Concepts in Gastric Intestinal Metaplasia and Gastric Cancer. Gastroenterol Hepatol (N Y). 2018 Feb;14(2):92-101. PMID 29606921
- [Background] Schulz C, Schutte K, Mayerle J, Malfertheiner P. The role of the gastric bacterial microbiome in gastric cancer: Helicobacter pylori and beyond. Therap Adv Gastroenterol. 2019 Dec 18;12:1756284819894062. doi: 10.1177/1756284819894062. eCollection 2019. PMID 31897087
- [Background] Cui J, Cui H, Yang M, Du S, Li J, Li Y, Liu L, Zhang X, Li S. Tongue coating microbiome as a potential biomarker for gastritis including precancerous cascade. Protein Cell. 2019 Jul;10(7):496-509. doi: 10.1007/s13238-018-0596-6. Epub 2018 Nov 26. PMID 30478535